CLINICAL TRIAL: NCT04819087
Title: Assessment Of The Effect Of Pelvic Floor Dysfunction Related Temporamandibular Joint Problems On Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Collaborators: MEDICANA HOSPITAL, ANKARA (Unknown)
Responsible Party: Principal Investigator, Nedim Uğur Kaya, LECTURER, KTO Karatay University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTOODY001
Record Dates: First submitted 2021-03-11; First posted 2021-03-26 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Tinnitus; Temporomandibular Joint Disorders; Pelvic Floor Disorders
Keywords: Tinnitus; Temporomandibular Joint Disorders; Pelvic Floor Disorders
MeSH Terms: conditions — Tinnitus; Temporomandibular Joint Disorders; Pelvic Floor Disorders | interventions — Surveys and Questionnaires; Biofeedback, Psychology; Electric Stimulation

STUDY DESIGN:
Intervention Model Description: It is planned to include patients diagnosed with pelvic floor dysfunction between the ages of 18-65 in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients (Experimental): Patients with Pelvic Floor Dysfunction Related Temporamandibular Joint Problems and Tinnitus
  Interventions: Behavioral: Questionnaires and Rehabilitation Programs

INTERVENTIONS:
Behavioral: Questionnaires and Rehabilitation Programs — Questionnaires and Rehabilitation Programs
  Other Names: Tinnitus Disability Questionnaire; Fonseca Questionnaire; Oral Habits Questionnaire; pelvic floor muscle rehabilitation with biofeedback; diaphragm breathing training; Electrical stimulation

SUMMARY:
The pelvic floor serves as stability and support as it is the postural balance and core resource base for the pelvic organs. A dysfunction in the organs in this area can affect the pelvic floor muscles, the functioning of an organs in the muscles. Incontinence organ prolapse, pelvic pain and sexual problems may occur when the support or stability of the pelvic floor is impaired. Pelvic floor novelization is not always seen weakness. Sometimes excessive contractions and excessive activity in muscle tone can be seen. Stress and anxiety-related tension are the main causes of pelvic floor dysfunctions. Involuntary contractions and excessive muscle tone in the pelvic floor muscles cause chronic pelvic pain syndrome, constipation and dyssynergic defecation problems. Some of these patients have complaints of tightening teeth in the temporamandibular joint, grinding teeth at night, together with contractions in the pelvic floor.

The aim of this study is to investigate the effect of pelvic floor improvement on tinnitus level as a result of dysfunctional condition in temporamandibular joint with treatment practices of pelvic floor patients with excessive muscle activity.

DETAILED DESCRIPTION:
The pelvic floor serves as stability and support as it is the postural balance and core resource base for the pelvic organs. A dysfunction in the organs in this area can affect the pelvic floor muscles, the functioning of an organs in the muscles. Incontinence organ prolapse, pelvic pain and sexual problems may occur when the support or stability of the pelvic floor is impaired. Pelvic floor novelization is not always seen weakness. Sometimes excessive contractions and excessive activity in muscle tone can be seen. Stress and anxiety-related tension are the main causes of pelvic floor dysfunctions. Involuntary contractions and excessive muscle tone in the pelvic floor muscles cause chronic pelvic pain syndrome, constipation and dyssynergic defecation problems. Some of these patients have complaints of tightening teeth in the temporamandibular joint, grinding teeth at night, together with contractions in the pelvic floor.

Diagnosis of patients in the temporamandibular joint is very difficult for the clinician. The difficulty of identifying etiological factors and the fact that dysfunction is associated with multifactorial factors make it mandatory to use different assessment methods in diagnosing patients with Temporamandibular joint dysfunction (TMD). One of the indexes used to diagnose TMD patients in a healthy population is the" Fonseca Anamnestic Index (FAI)". The low cost and easy applicability of the index make it preferred for TMD patients at the stage of diagnosis (Ayalı ve Ramoğlu, 2014; Türken vd., 2020).

In the pathogenesis of TMD, parafunctional habits such as day and night tooth tightening, tooth grinding, nail eating, lip biting, cheek biting, pen biting, chewing gum play an important role. It has been reported that there is often a positive correlation between TMD and parafunctional habits. "Oral Behavior Checklist (OBC)" is used in the diagnosis of such oral habits (Güngör, 2019; Türken vd., 2020).

It is thought that this dysfunctional condition in the temporamandibular joint may cause tinnitus in patients. The fact that tinnitus is subjective and an unsolved symptom related to the mechanisms of its occurrence makes it difficult to obtain objective assessment and concrete data. For this reason, the evaluation of tinnitus is again possible by perceptual measurement. For this purpose, psychoacoustic tests such as tinnitus intensity and frequency matching, maskability, residual inhibition, and verbal, numerical, and visual rating scales are used to evaluate tinnitus (Meikle vd., 2008). The Tinnitus Disability Questionnaire is the only scale with validity and reliability in Turkish and is widely used in our country to determine the level of tinnitus (Aksoy vd., 2007).

Although the use of scale is an important tool in determining the level of tinnitus, it is difficult for each person to express their condition as it is. It is known that some patients may exaggerate or underestimate their complaints, each scale has strengths and weaknesses, and sensitivity may vary depending on the therapy used. Since most of the scales are developed in English, it should be considered that when applied to different cultures and socio-economic groups, there may be changes in specificity and sensitivity (Langguth vd., 2006). For this reason, the addition of a structured interview form as a standard in addition to the scale strengthens the opinion of the clinician.

Accordingly, it is expected that temporamandibular joint loosens after treatment applications in patients with pelvic floor dysfunction. As a result of this relaxation, we believe that there may be a decrease in the level of tinnitus felt in patients.

The aim of this study is to investigate the effect of pelvic floor improvement on tinnitus level as a result of dysfunctional condition in temporamandibular joint with treatment practices of pelvic floor patients with excessive muscle activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-65 years
* Patients with Pelvic Plate Disorders
* Patients with Tinnitus Patients with Temporomandibular Joint Disorders

Exclusion Criteria:

* Patients under 18 years and over 65 years
* Patients without Pelvic Plate Disorders
* Patients without Tinnitus
* Patients without Temporomandibular Joint Disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Tinnitus Disability Questionnaire | Change from Baseline and 10 Weeks
  The application of the questionnaire, which is not affected by hearing loss, age and gender, gives both easy and psychometric clearer measurements. The questionnaire consisting of 25 questions examines the perception of tinnitus and psychosocial status of the patient
Fonseca Anamnestic Index | Change from Baseline and 10 Weeks
  FAI is a questionnaire consisting of 10 questions that determine the presence of pain in TME, head, back areas and during chewing, parafunctional habits, movement restriction, clique, malocclusion, emotional stress
Oral Behavioral Survey Questions | Change from Baseline and 10 Weeks
  In the pathogenesis of TMD, parafunctional habits such as day and night tooth tightening, tooth grinding, nail eating, lip biting, cheek biting, pen biting, chewing gum play an important role. A positive association has often been reported between TMD and parafunctional habits. "Oral Behavior Checklist (OBC)", a survey study consisting of 21 Questions, is used to diagnose such oral habits

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay Üniversitesi, Konya, Karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aksoy S, Firat Y, Alpar R. The Tinnitus Handicap Inventory: a study of validity and reliability. Int Tinnitus J. 2007;13(2):94-8. PMID 18229787
- [Background] Ayalı, A., Ramoğlu, S. (2014). Kuzey kıbrıs'ta diş hekimliği fakültesi öğrencilerinde temporomandibuler eklem disfonksiyonu'nun prevalansı ve şiddetinin araştırılması, Atatürk Üniv. Diş Hek. Fak. Derg. Cilt:24, Sayı:3, Yıl: 2014, Sayfa: 367-372
- [Background] Langguth B, Goodey R, Azevedo A, Bjorne A, Cacace A, Crocetti A, Del Bo L, De Ridder D, Diges I, Elbert T, Flor H, Herraiz C, Ganz Sanchez T, Eichhammer P, Figueiredo R, Hajak G, Kleinjung T, Landgrebe M, Londero A, Lainez MJ, Mazzoli M, Meikle MB, Melcher J, Rauschecker JP, Sand PG, Struve M, Van de Heyning P, Van Dijk P, Vergara R. Consensus for tinnitus patient assessment and treatment outcome measurement: Tinnitus Research Initiative meeting, Regensburg, July 2006. Prog Brain Res. 2007;166:525-36. doi: 10.1016/S0079-6123(07)66050-6. PMID 17956816
- [Background] Türken, R., Büyük, S. K., Yaşa, Y. (2020). Diş Hekimliği Fakültesi Öğrencilerinde Temporomandibular Eklem Rahatsızlıklarının ve Ağız Sağlığı Alışkanlıklarının Değerlendirilmesi, ACU Sağlık Bil Derg 2020; 11(2):208-213, https://doi.org/10.31067/0.2018.83